CLINICAL TRIAL: NCT05474911
Title: RANDOMIZED COMPARATIVE CLINICAL STUDY BETWEEN TWO TREATMENT STRATEGIES IN PATIENTS WITH PILONIDAL SINUS: CONVENTIONAL CARE VERSUS NEGATIVE PRESSURE THERAPY.
Brief Title: PILONIDAL SINUS: CONVENTIONAL CARE VERSUS NEGATIVE PRESSURE THERAPY.
Acronym: SINUS-TPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sebastiano Biondo (Other)
Collaborators: Hospital Universitari de Bellvitge (Other)
Responsible Party: Sponsor-Investigator, Sebastiano Biondo, PhD, MD, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICPS020/22
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Pilonidal Sinus; Wound Heal
Keywords: Negative presure therapy
MeSH Terms: conditions — Pilonidal Sinus | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional care (Active Comparator)
  Interventions: Other: Conventional wound care
- Negative pressure therapy (Experimental)
  Interventions: Device: Negative pressure therapy

INTERVENTIONS:
Device: Negative pressure therapy — The wound will be cleaned (irrigation with Physiological Serum), the cavity and the perilesional area will be dried with gauze. A skin protection spray will be applied to avoid irritation of the skin around the wound due to the adhesive of the dressing. The cavity will be filled with a sponge. When the depth of the wound is less than 1.5 cm, it will not be necessary to fill the defect. The appropriate dressing will be applied to the size of the incision, reinforcing the edges, and it will be connected to the TPN device, ensuring correct functionality.
  Arms: Negative pressure therapy
Other: Conventional wound care — The wound will be cleaned with physiological serum irrigation, the cavity will be dried with gauzes and filled with a dressing made of cellulose and silver. A skin protection spray will be applied to avoid irritation of the skin around the wound due to the adhesive of the dressing.
  Arms: Conventional care

SUMMARY:
Pilonidal Sinus PS is a prevalent disease in young patients. There is currently no consensus on the surgical treatment of choice. Each method is associated with different advantages and disadvantages, as well as different recurrence rates. The ideal treatment should reduce morbidity, be associated with a short hospital stay (outpatient surgery), promote rapid healing, early return to work, and have a low recurrence rate. To date, no technique meets all these criteria. However, the NPT could meet them. The use of NPT in PS could decrease healing time, achieving an early return to work. In addition, it would avoid the need for daily dressings, which would mean lower hospital costs. However, the location of the wound (sacrum) and its proximity to the anal margin mean that its use cannot be generalized.

Although two retrospective series have recently reported good results with the use of NPT in PS, a prospective, randomized study is needed to compare healing time, recurrence rates, hospital costs, and assess quality of life for determine if this could be the treatment of choice.

Although NPT is commonly used in clinical practice (being useful in closing complex wounds, with devitalized tissues, burns and wounds with exposed tendons), to date there is not enough evidence to support its use after flattening the PS and it is for this reason that we conducted this study.

In this project there is a total absence of commercial interest in the proposal. No project related to the proposed one is currently being carried out.

DETAILED DESCRIPTION:
The study population will be made up of all patients with PS admitted to the General and Digestive Surgery service of the Hospital Universitari de Bellvitge from the start of the trial until the end of recruitment, and who meet the inclusion criteria.

Once the patients belonging to the population of interest have been identified, they will propose to participate in the clinical trial, providing complete information, as well as an information sheet with the details of the study. If you agree, the informed consent document will be provided for your signature and randomization will proceed.

Bitter et al. observed in a prospective study that the use of NTP did not reduce healing time compared to conventional closure 84 days (34-349) vs 93 days (43-264); p=0.44. However, the duration of NPT application of only 2 weeks might have been too short to see an adequate effect. Also, the small sample size could have influenced the results. On the other hand, recent publications on the use of TPN in the treatment of pilonidal sinus have shown a significant reduction in healing time (28 days) with minimal complications and adequate patient satisfaction. Taking into account the scarce evidence of the studies cited, we have decided to adopt a conservative criterion, assuming a smaller difference in time to healing between the two treatments (35 days).

To calculate the sample size, the time variable has been transformed into a logarithm. Accepting an alpha risk of 0.05 and a beta risk of 0.20 in a bilateral contrast, 94 patients, 47 subjects in the control group and 47 in the experimental group, are needed to detect a difference of 0.77. A common standard deviation of 1.26 is assumed. A rate of loss to follow-up of 10% has been estimated.

Randomization 1:1 will be performed using a statistical program at the baseline visit in outpatient clinics 48 hours after surgery, after assessing the dimensions of the wound, checking whether the participant meets the inclusion/exclusion criteria and has signed the informed consent.

For the purposes of the study and in order not to influence the type of surgery performed on patients with PS, only those patients who have undergone a flattening will be included. The 1st cure will be performed 24 hours later in the area outpatient clinic and will consist of removing the dressing, washing with physiological serum and placing a dry dressing.

48 hours after surgery, patients will be evaluated in outpatient clinics at our hospital. The dressing will be removed from the wound and after washing with serum, it will be checked if the patient meets the inclusion criteria. If you meet them, you will be offered to participate in the study and once you have signed the informed consent, randomization will proceed.

The patients will be monitored in person in outpatient clinics (CEX) by two members of the research team, made up of a nurse specialized in cures and a doctor specialized in surgery.

During the follow-up visits, a conventional dressing will be performed or the negative pressure system will be changed. Symptomatology and quality of life data will be collected through validated surveys.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with SP (recurrence or not), who have undergone surgery.
* Minimum depth of the wound 1.5 cm.

Exclusion Criteria:

* Inferior margin of the surgical wound is located less than 3 cm from the anus
* Patients under 16 years of age
* Unable to track
* Diagnosed psychiatric illness
* Patients diagnosed with hidradenitis
* Uncontrolled diabetics
* Immunocompromised (kidney or liver transplant, chronic treatment with corticosteroids, haematological disease, neoplastic disease undergoing chemotherapy)

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Cicatrization | 1 year
  Time in days from surgery to complete epithelialization of the wound, assessed by the dressing nurse and surgeon.

SECONDARY OUTCOMES:
Wound size | 1 year
  Defined as wound volume measured in milliliters. In addition, the measurements of width, length and depth in cm will be collected.
Postoperative pain | 1 year
  Evaluated with the visual analog pain scale ranging from 0 to 10, where 0 represents no pain and 10 represents intolerable pain. It will be assessed weekly
Time of incorporation into daily activities | 1 year
  Time in days from surgery to incorporation into daily activities as reported by the patients in the weekly evaluation
Patient quality of life | 1 year
  Evaluated by applying the SF-36 questionnaire in both groups at 15 days, 30 days, and monthly until healing. A total score will be calculated in each of the 8 sections and converted to a scale from 0 to 100, with a score of 0 equivalent to maximum disability and a score of 100 equivalent to no disability.
Patient satisfaction | 1 year
  Reported by the patient on a scale of 0 to 10, where 0 corresponds to "totally unsatisfactory" and 10 corresponds to "totally satisfactory". The score obtained at the end of healing will be recorded. It will be done when healing is complete.
Adverse effects related to the treatments | 1 year
  Reported adverse effects
Cost effectiveness | 1 year
  Cost effectiveness of NPT
Disease recurrence at follow-up | 1 year
  Disease recurrence will be assessed 1 year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Biondo, MD, Study Chair — Hospital Universitari de Bellvitge
Locations (1):
- Bellvitge University Hospital, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roldon Golet M, Siles Hinojosa A, Gonzalez Ruiz Y, Escartin Villacampa R, Goded Broto I, Bragagnini Rodriguez P. Pilonidal sinus in adolescence: is there an ideal surgical approach? Cir Pediatr. 2021 Jul 1;34(3):119-124. English, Spanish. PMID 34254748
- [Background] Kumar M, Clay WH, Lee MJ, Brown SR, Hind D. A mapping review of sacrococcygeal pilonidal sinus disease. Tech Coloproctol. 2021 Jun;25(6):675-682. doi: 10.1007/s10151-021-02432-9. Epub 2021 Mar 16. PMID 33728570
- [Background] Caliskan M, Kosmaz K, Subasi IE, Acar A, Evren I, Bas G, Atayoglu AT. Comparison of Common Surgical Procedures in Non-complicated Pilonidal Sinus Disease, a 7-Year Follow-Up Trial. World J Surg. 2020 Apr;44(4):1091-1098. doi: 10.1007/s00268-019-05331-1. PMID 31848678
- [Background] Luedi MM, Schober P, Stauffer VK, Diekmann M, Andereggen L, Doll D. Gender-specific prevalence of pilonidal sinus disease over time: A systematic review and meta-analysis. ANZ J Surg. 2021 Jul;91(7-8):1582-1587. doi: 10.1111/ans.16990. Epub 2021 Jun 7. PMID 34101331
- [Background] Bi S, Sun K, Chen S, Gu J. Surgical procedures in the pilonidal sinus disease: a systematic review and network meta-analysis. Sci Rep. 2020 Aug 13;10(1):13720. doi: 10.1038/s41598-020-70641-7. PMID 32792519
- [Background] Al-Khamis A, McCallum I, King PM, Bruce J. Healing by primary versus secondary intention after surgical treatment for pilonidal sinus. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD006213. doi: 10.1002/14651858.CD006213.pub3. PMID 20091589
- [Background] Grabowski J, Oyetunji TA, Goldin AB, Baird R, Gosain A, Lal DR, Kawaguchi A, Downard C, Sola JE, Arthur LG, Shelton J, Diefenbach KA, Kelley-Quon LI, Williams RF, Ricca RL, Dasgupta R, St Peter SD, Somme S, Guner YS, Jancelewicz T. The management of pilonidal disease: A systematic review. J Pediatr Surg. 2019 Nov;54(11):2210-2221. doi: 10.1016/j.jpedsurg.2019.02.055. Epub 2019 Mar 19. PMID 30948198
- [Background] Iesalnieks I, Ommer A, Petersen S, Doll D, Herold A. German national guideline on the management of pilonidal disease. Langenbecks Arch Surg. 2016 Aug;401(5):599-609. doi: 10.1007/s00423-016-1463-7. Epub 2016 Jun 16. PMID 27311698
- [Background] Stauffer VK, Luedi MM, Kauf P, Schmid M, Diekmann M, Wieferich K, Schnuriger B, Doll D. Common surgical procedures in pilonidal sinus disease: A meta-analysis, merged data analysis, and comprehensive study on recurrence. Sci Rep. 2018 Feb 15;8(1):3058. doi: 10.1038/s41598-018-20143-4. PMID 29449548
- [Background] McCallum IJ, King PM, Bruce J. Healing by primary closure versus open healing after surgery for pilonidal sinus: systematic review and meta-analysis. BMJ. 2008 Apr 19;336(7649):868-71. doi: 10.1136/bmj.39517.808160.BE. Epub 2008 Apr 7. PMID 18390914
- [Background] Johnson EK, Vogel JD, Cowan ML, Feingold DL, Steele SR; Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons' Clinical Practice Guidelines for the Management of Pilonidal Disease. Dis Colon Rectum. 2019 Feb;62(2):146-157. doi: 10.1097/DCR.0000000000001237. No abstract available. PMID 30640830
- [Background] Calisir A, Ece I. Comparison of the Keystone flap and the Limberg flap technique in the surgical treatment of pilonidal sinus disease. Updates Surg. 2021 Dec;73(6):2341-2346. doi: 10.1007/s13304-021-01153-w. Epub 2021 Aug 20. PMID 34417712
- [Background] Prassas D, Rolfs TM, Schumacher FJ, Krieg A. Karydakis flap reconstruction versus Limberg flap transposition for pilonidal sinus disease: a meta-analysis of randomized controlled trials. Langenbecks Arch Surg. 2018 Aug;403(5):547-554. doi: 10.1007/s00423-018-1697-7. Epub 2018 Jul 31. PMID 30066108
- [Background] Maranna H, Lal P, Mishra A, Bains L, Sawant G, Bhatia R, Kumar P, Beg MY. Negative pressure wound therapy in grade 1 and 2 diabetic foot ulcers: A randomized controlled study. Diabetes Metab Syndr. 2021 Jan-Feb;15(1):365-371. doi: 10.1016/j.dsx.2021.01.014. Epub 2021 Jan 23. PMID 33524646
- [Background] Liu Z, Dumville JC, Hinchliffe RJ, Cullum N, Game F, Stubbs N, Sweeting M, Peinemann F. Negative pressure wound therapy for treating foot wounds in people with diabetes mellitus. Cochrane Database Syst Rev. 2018 Oct 17;10(10):CD010318. doi: 10.1002/14651858.CD010318.pub3. PMID 30328611
- [Background] Kojima K, Goto M, Nagashima Y, Saito Y, Kawai M, Takebe S, Egawa A, Tanba M, Ishikawa K, Matsuoka H, Masaki T, Sunami E, Ohura N, Teruya K, Eto K, Nozawa K, Sakamoto K, Funahashi K. Effectiveness of negative pressure wound therapy for the wound of ileostomy closure: a multicenter, phase II randomized controlled trial. BMC Surg. 2021 Dec 28;21(1):442. doi: 10.1186/s12893-021-01446-2. PMID 34963451
- [Background] Chen L, Zhang S, Da J, Wu W, Ma F, Tang C, Li G, Zhong D, Liao B. A systematic review and meta-analysis of efficacy and safety of negative pressure wound therapy in the treatment of diabetic foot ulcer. Ann Palliat Med. 2021 Oct;10(10):10830-10839. doi: 10.21037/apm-21-2476. PMID 34763444
- [Background] Hyldig N, Birke-Sorensen H, Kruse M, Vinter C, Joergensen JS, Sorensen JA, Mogensen O, Lamont RF, Bille C. Meta-analysis of negative-pressure wound therapy for closed surgical incisions. Br J Surg. 2016 Apr;103(5):477-86. doi: 10.1002/bjs.10084. PMID 26994715
- [Background] Searle RJ, Myers D. A survey of caesarean section surgical site infections with PICO Single Use Negative Pressure Wound Therapy System in high-risk patients in England and Ireland. J Hosp Infect. 2017 Oct;97(2):122-124. doi: 10.1016/j.jhin.2017.02.023. Epub 2017 Aug 12. PMID 28807639
- [Background] Meyer J, Roos E, Abbassi Z, Buchs NC, Ris F, Toso C. Prophylactic Negative-pressure Wound Therapy Prevents Surgical Site Infection in Abdominal Surgery: An Updated Systematic Review and Meta-analysis of Randomized Controlled Trials and Observational Studies. Clin Infect Dis. 2021 Dec 6;73(11):e3804-e3813. doi: 10.1093/cid/ciaa1203. PMID 32818259
- [Background] Frear CC, Griffin BR, Cuttle L, Kimble RM, McPhail SM. Cost-effectiveness of adjunctive negative pressure wound therapy in paediatric burn care: evidence from the SONATA in C randomised controlled trial. Sci Rep. 2021 Aug 17;11(1):16650. doi: 10.1038/s41598-021-95893-9. PMID 34404842
- [Background] Saunders C, Nherera LM, Horner A, Trueman P. Single-use negative-pressure wound therapy versus conventional dressings for closed surgical incisions: systematic literature review and meta-analysis. BJS Open. 2021 Jan 8;5(1):zraa003. doi: 10.1093/bjsopen/zraa003. PMID 33609382
- [Background] Cheung DC, Muaddi H, de Almeida JR, Finelli A, Karanicolas P. Cost-Effectiveness Analysis of Negative Pressure Wound Therapy to Prevent Surgical Site Infection After Elective Colorectal Surgery. Dis Colon Rectum. 2022 May 1;65(5):767-776. doi: 10.1097/DCR.0000000000002154. PMID 34840300
- [Background] Berner-Hansen V, Oma E, Willaume M, Jensen KK. Prophylactic negative pressure wound therapy after open ventral hernia repair: a systematic review and meta-analysis. Hernia. 2021 Dec;25(6):1481-1490. doi: 10.1007/s10029-021-02485-7. Epub 2021 Aug 14. PMID 34392436
- [Background] Gao J, Wang Y, Song J, Li Z, Ren J, Wang P. Negative pressure wound therapy for surgical site infections: A systematic review and meta-analysis. J Adv Nurs. 2021 Oct;77(10):3980-3990. doi: 10.1111/jan.14876. Epub 2021 Apr 27. PMID 33905552
- [Background] Payne C, Edwards D. Application of the Single Use Negative Pressure Wound Therapy Device (PICO) on a Heterogeneous Group of Surgical and Traumatic Wounds. Eplasty. 2014 Apr 28;14:e20. eCollection 2014. PMID 24917894
- [Background] Kim S, Kang SI. The effectiveness of negative-pressure wound therapy for wound healing after stoma reversal: a randomised control study (SR-PICO study). Trials. 2020 Jan 6;21(1):24. doi: 10.1186/s13063-019-3925-z. PMID 31907033
- [Background] Milone M, Basso L, Manigrasso M, Pietroletti R, Bondurri A, La Torre M, Milito G, Pozzo M, Segre D, Perinotti R, Gallo G. Consensus statement of the Italian society of colorectal surgery (SICCR): management and treatment of pilonidal disease. Tech Coloproctol. 2021 Dec;25(12):1269-1280. doi: 10.1007/s10151-021-02487-8. Epub 2021 Jun 27. PMID 34176001
- [Background] Hannan E, Harding T, Feizal H, Martin S. Negative pressure wound therapy following excision of pilonidal sinus disease: A retrospective review. Colorectal Dis. 2021 Nov;23(11):2961-2966. doi: 10.1111/codi.15890. Epub 2021 Sep 12. PMID 34455675
- [Background] Giordano P, Schembari E, Keshishian K, Leo CA. Negative pressure-assisted endoscopic pilonidal sinus treatment. Tech Coloproctol. 2021 Jun;25(6):739-743. doi: 10.1007/s10151-021-02431-w. Epub 2021 Mar 23. PMID 33755853